CLINICAL TRIAL: NCT01497301
Title: Initiating Diabetic Group Visits in Newly Diagnosed Diabetics in an Urban Academic Medical Practice
Brief Title: Efficacy Study of Diabetes Group Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Holly Hofkamp, Clinical Instructor, Department of Family Medicine, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00007909
Record Dates: First submitted 2011-12-19; First posted 2011-12-22 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Group Visit; Shared Medical Appointment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Individual Medical Appointment (No Intervention)
- Group Visits (Active Comparator)
  Interventions: Behavioral: Group Visits

INTERVENTIONS:
Behavioral: Group Visits — During group visits, there will be discussions regarding the basic pathophysiology of diabetes, the "ABCs to Better Diabetic Care" as defined by the ACP Diabetes Care Guide, setting goals, nutrition, exercise, diabetic medications, and complications of diabetes. Patients will have blood drawn to measure hemoglobin A1C and lipids. They will be educated on self glucose monitoring so they will undergo finger sticks to measure their own glucose. BP measurements, monofilament foot exams, and urine collection for microalbumin will also occur during the study. They may also receive immunizations. A consent form for participation in the group visits, including undergoing the above procedures will be reviewed at our first group visit and signed by all participants.
  Arms: Group Visits

SUMMARY:
Much evidence exists that new, more effective methods of delivering care to diabetics are necessary. In our current system of delivering care, diabetes care is often done in the context of multiple other issues addressed during a regular office visit. Providers often lack the time to properly educate patients on diabetes self management topics. This project hopes to show that group visits can improve clinical outcomes, patient satisfaction, provider satisfaction, and patient's self management knowledge, while decreasing cost. This group visit method can make care more patient-centered and team based which is in alignment with our organization's goal of becoming a true patient centered medical home. If successful, this could expand to our other family medicine clinic sites and provide a valuable learning opportunity for the family medicine residents at OHSU.

The investigators will first identify newly diagnosed diabetics (diagnosed within the last 12 months) at the South Waterfront and Gabriel Park family medicine clinics using EPIC. The investigators will invite those diabetics identified from the South Waterfront clinic to participate in 6 group visits that will follow a curriculum that the investigators created based on the National Standards for Diabetes Self Management Education and the ACP Diabetes Care Guide. This curriculum will address basic pathophysiology of diabetes, the "ABCs to Better Diabetic Care" as defined by the ACP Diabetes Care Guide, setting goals, nutrition, exercise, diabetic medications, and complications of diabetes. This intervention group will be compared to a control cohort identified at the Gabriel Park clinic that will continue to receive standard diabetes care from their primary physician. The investigators will look at and compare clinical outcomes (Hemoglobin A1C, blood pressure (BP), and LDL cholesterol levels), adherence to recommended preventive measures for diabetics (foot exams, eye exams, yearly microalbumin, and immunizations), patient and provider satisfaction, as well as cost. Cost data will be collected using EPIC to look at the costs involved in group visits compared to the cost of delivering diabetic care through the standard individual medical appointment. The investigators may also use EPIC to look at utilization of specialty services, emergency room visits, and inpatient admissions and compared utilization across groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus, type 2 after 11/01/2010
* English speaking

Exclusion Criteria:

* Dementia
* Unable to come to all 6 preschedule group visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C | baseline, 6 months, and 12 months

SECONDARY OUTCOMES:
Number of patients that are in compliance with all recommended preventive measures for diabetics | baseline, 6 months, and 12 months
  Recommended preventive measures for diabetics include yearly foot exams, yearly eye exams, yearly microalbumin. This also includes yearly immunization with influenza vaccine and immunization with pneumococcal vaccine once before age 65 and once after age 65.
Patient satisfaction with diabetes group visits | 6 months and 12 months
  Will use validated tool: Diabetes Management Evaluation Tool
Provider Satisfaction with Diabetes Group Visits | baseline, 6 months, 12 months
Difference in costs of delivering care to diabetics through group visits compared to standard individual medical appointments | 6 months, 12 months
Change in blood pressure | baseline, 6 months, 12 months
Change in LDL cholesterol | baseline, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Scott Fields, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States